CLINICAL TRIAL: NCT02587156
Title: Fate of Nutrient-Derived Amino Acids: Influence of Habituated Levels of Daily Dietary Protein Intake on Protein Utilization
Brief Title: Fate of Nutrient-Derived Amino Acids, FONDAA
Acronym: FONDAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Grith Højfeldt, MSc. Human Biology - PhD student, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBH122
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Protein Utilization; Dietary Protein
Keywords: Required dietary protein; Amino acid; Splanchnic extraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meal serving at high dietary protein (Experimental): Test the handling of meal-served protein when habituated to high dietary protein at an amount above 1.5 g protein/kg/day
  Interventions: Dietary Supplement: Meal serving at high dietary protein; Dietary Supplement: Meal serving
- Meal serving at low dietary protein (Active Comparator): Test the handling of meal-served protein when habituated to high dietary protein at an amount below 0.8 g protein/kg/day
  Interventions: Dietary Supplement: Meal serving at low dietary protein; Dietary Supplement: Meal serving

INTERVENTIONS:
Dietary Supplement: Meal serving at high dietary protein — Participants are habituated to a high level of dietary protein intake for 21 days.
  Arms: Meal serving at high dietary protein
Dietary Supplement: Meal serving at low dietary protein — Participants are habituated to a low level of dietary protein intake for 21 days.
  Arms: Meal serving at low dietary protein
Dietary Supplement: Meal serving — To investigate impact of habituated protein level

SUMMARY:
12 elderly (65-70 years of age) male subjects will be included and complete a double blinded cross-over study. They will be habituated for 21 days to either low or high protein intake (below 0.8 g/kg or above 1.5 g/kg, respectively). Following a 45 day washout period they will switch to the alternate group. At the end of each habituation period, the investigators will measure the appearance of labelled amino acids from milk proteins.

ELIGIBILITY:
Exclusion Criteria:

* Hyperlipidemia
* Hypertension

Inclusion Criteria:

* Males age 65-70
* Independently dwelling
* Without any major health issues (blood pressure, cholesterol and lipid profile will be measured and evaluated by a physician)
* Non-diabetic
* No organ disease
* No back pain
* Not regularly take any prescription drugs or dietary supplements, which can influence muscle protein synthesis
* Alcohol intake below 21 units pr. week
* No known arthrosclerosis

Ages: 65 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Abundance of milk protein-bound amino acid labels in blood protein. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  After intake of milk proteins at time 0 (zero) the quantity of intrinsic labels D5-phe from whey and 15N-phe from casein will be measured in liver-synthesized blood protein at 240 min.

SECONDARY OUTCOMES:
Abundance of milk protein-bound amino acid labels in myofibrillar protein. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  After intake of milk proteins at time 0 (zero) the quantity of intrinsic labels D5-phe from whey and 15N-phe from casein will be measured in myofibrillar protein at 240 min.
Leg phenylalanine rate of disappearance and appearance, net balance. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From arterial and femoral venous blood samples obtained at baseline, 30, 60, 90, 120, 150, 180, 240 min phenylalanine tracer enrichments and concentrations as well as plasma flow will be measured.
First pass splanchnic extraction of dietary protein-derived labeled phenylalanine. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From hepatic venous blood samples obtained at baseline, 30, 60, 90, 120, 150, 180, 240 min phenylalanine tracer enrichments and concentrations as well as plasma flow will be measured. Knowing the amount of ingested protein and labeled phenylalanine we can calculate the first pass splanchnic amino acid extraction.
Whole body phenylalanine rate of disappearance and appearance, net balance. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From blood samples obtained at baseline, 30, 60, 90, 120, 150, 180, 240 min phenylalanine tracer enrichments will be measured.
The myofibrillar protein fractional synthesis rate | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From muscle biopsies obtained at baseline, 60 and 240 min the abundance of phenylalanine tracer bound in the myofibrillar proteins will be measured and the fractional synthesis rate will be measured within the first from baseline to 60 min and 240 min as well as from 60-240 min postprandial.
Response of expression of proteins involved in muscle protein turnover | Baseline, 60 min and 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From baseline to 60 and 240 min after intake of the standardized meal after 21 days of habituation to either a high or a low dietary protein intake expression of signalling proteins related to protein turnover in the muscle will be measured by use of western blotting.
Urea production. | Baseline to 240 min postprandial
  Related to the trials conducted after 21 days of habituation to either high or low protein in the diet:
  From blood samples obtained at baseline, 30, 60, 90, 120, 150, 180, 240 min urea tracer enrichments and concentrations will be measured. With this, and flow measurements, we can determine the rate of urea production.
Nitrogen and creatinine excreted in urine | 21 days post intervention, 240 min postprandial and 24 hours post the day 21 trial day
  Related to the adaptation to the 21 day habituation period to either high or low protein in the diet as well as the response to the standardized trial meal:
  Nitrogen and creatinine content is measured in urine is collected for the last 24 h of the 21 day habituation period, as well as during the 240 min trial day and the remaining 20 hours of the trial day.
Fecal microbiota composition | Change from pre-intervention to 21 days and 22 days (21 intervention days habituation and the standardized trial meal on day 21)
  Related to the adaptation to the 21 day habituation period to either high or low protein in the diet as well as the response to the standardized trial meal:
  The microbiota compositions, will be measured in fecal samples collected before the 21 day habituation period, after the 21 day habituation periode, as well as after the 240 min trial day
Adaptation of expression of proteins involved in muscle protein turnover | After 21 days of habituation to either a high or a low dietary protein intake.
  Related to the adaptation to the 21 day habituation period to either high or low protein in the diet:
  Biopsies taken following the two 21 day habituation period will, by use of western blotting, be analysed for expression of signalling proteins involved in muscle protein turnover.

CONTACTS AND LOCATIONS:
Overall Officials: Grith Højfeldt, M.Sc., Principal Investigator — Bispebjerg Hospital; Lars Holm, Ph.D., Principal Investigator — Bispebjerg Hospital
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hojfeldt G, Bulow J, Agergaard J, Asmar A, Schjerling P, Simonsen L, Bulow J, van Hall G, Holm L. Impact of habituated dietary protein intake on fasting and postprandial whole-body protein turnover and splanchnic amino acid metabolism in elderly men: a randomized, controlled, crossover trial. Am J Clin Nutr. 2020 Dec 10;112(6):1468-1484. doi: 10.1093/ajcn/nqaa201. PMID 32710741